CLINICAL TRIAL: NCT01597297
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Exploratory Study to Assess the Effect of Treatment With Prolonged-Release Fampridine (BIIB041) 10 mg Twice Daily on Walking Ability and Balance in Subjects With Multiple Sclerosis
Brief Title: Exploratory Study to Assess the Effect of Fampridine (BIIB041) on Walking Ability and Balance in Participants With Multiple Sclerosis.
Acronym: MOBILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 218MS205; 2012-000368-90
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fampridine-PR (Experimental): Prolonged-Release Fampridine (Fampridine-PR) 10 mg twice daily (every 12 hours) for up to 24 weeks.
  Interventions: Drug: BIIB041 (PR Fampridine)
- Placebo (Placebo Comparator): Matched placebo twice daily (every 12 hours) for up to 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BIIB041 (PR Fampridine) — 10 mg twice daily, given orally. Doses of study treatment must be spaced at least 12 hours apart. If a dose of study treatment is delayed or missed, the participant should not dose again until their next scheduled dose. Tablets must be swallowed whole and should be taken without food.
  Other Names: Fampridine-PR (prolonged-release); Dalfampridine-ER (extended-release); FAMPYRA®; AMPYRA®
  Arms: Fampridine-PR
Other: Placebo — Twice daily, given orally. Doses of study treatment must be spaced at least 12 hours apart. If a dose of study treatment is delayed or missed, the participant should not dose again until their next scheduled dose. Tablets must be swallowed whole and should be taken without food.
  Arms: Placebo

SUMMARY:
The objectives of this study in Multiple Sclerosis (MS) participants treated with prolonged-released fampridine (BIIB041) 10 mg twice daily compared with participants treated with placebo are to assess the effect over 24 weeks on the following parameters to explore endpoints for the Phase 3 study: self-assessed walking disability, dynamic and static balance, subjective impression of well-being, and participants' global impression of change in walking . Another purpose of this study is to evaluate the safety and tolerability of prolonged-release fampridine.

DETAILED DESCRIPTION:
The primary objective of the study is to explore the effect of prolonged-released fampridine 10 mg twice daily in patients with Multiple Sclerosis with walking disability. The change of walking ability will be measured using Multiple Sclerosis Walking Scale-12 (MSWS-12) to further elucidate the clinical relevance of changes over 24 weeks treatment duration. Another purpose of this study is to evaluate the safety and tolerability of prolonged-release fampridine.

Approximately 120 patients MS will be randomized over 20 sites worldwide. Duration of patient's participation in the study will be approximately 28 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be able to understand the purpose and risk of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations
* Diagnosis of primary-progressive, secondary progressive, progressive-remitting, or relapsing-remitting Multiple Sclerosis of at least 3-month duration
* EDSS 4 to 7
* Female patients of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment
* Must be able to understand and comply with the requirements of the protocol

Key Exclusion Criteria:

* Known allergy to pyridine-containing substances or to any of the inactive ingredients in the prolonged release fampridine (BIIB041) tablet
* Any history of seizure, epilepsy, or other convulsive disorder, with the exception of febrile seizures in childhood
* An estimated creatinine clearance (CrCl) of <80 mL/minute (using the Cockcroft-Gault formula)
* Known history of Human Immunodeficiency Virus, hepatitis C, or hepatitis B. Subjects who have evidence of prior hepatitis infection that has been serologically confirmed as resolved based on previous testing documented in the subjects' medical history are not excluded from study participation
* History of malignant disease including solid tumors and hematologic malignancies (with the exception of basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured) within the 5 years prior to the Screening Visit, or at any time during the screening period
* Onset of MS exacerbation within the 60 days prior to the Screening Visit, or at any time during the screening period
* History of any major surgical intervention (with the exception of skin biopsy) within the 30 days prior to the Screening Visit, or at any time during the screening period
* Any non-MS-related condition or factor (as determined by the Investigator) that is likely to interfere with walking ability including, but not limited to, previous major surgery of the foot, leg, or hip; any significant trauma; or known peripheral neuropathy of the lower limb
* Presence of pulmonary disease including, but not limited to, chronic obstructive pulmonary disease that could impede the subject's daily activities (as determined by the Investigator)
* Presence of any psychiatric disorder, including clinical depression, that is likely to interfere with the subject's participation in the study (as determined by the Investigator)
* Uncontrolled hypertension (as determined by the Investigator) at the Screening Visit, any time during the screening period, or Day 1
* History of any clinically significant endocrinologic, hematologic, immunologic, metabolic, urologic, neurologic (except for MS, but including events indicative of a potentially lower seizure threshold), dermatologic, or other major disease (as determined by the Investigator)
* Clinically significant abnormal laboratory values (as determined by the Investigator)
* A Body Mass Index ≥40
* Use of off label MS treatment including rituximab, alemtuzumab, daclizumab, or antibody (except natalizumab) within the 3 months prior to the Screening Visit, or any time during the screening period, or scheduled use during study participation
* Use of mitoxantrone or cyclophosphamide within the 3 months prior to the Screening Visit, or any time during the screening period, or scheduled use during study participation
* Initiation of natalizumab treatment or any change in the subject's dose or regimen of natalizumab, within the 3 months prior to the Screening Visit, or at any time during the screening period
* Initiation of treatment with, or any change in the subject's dose or regimen of, interferon β 1b, interferon β-1a, fingolimod, or glatiramer acetate within the 30 days prior to the Screening Visit, or at any time during the screening period
* Pulsed steroid treatment within the 60 days prior to the Screening Visit, or at any time during the screening period
* Any change in the subject's medication dose or regimen for the treatment of fatigue or depression within the 30 days prior to the Screening Visit, or at any time during the screening period
* Any change in prophylactic treatment for pain with antidepressants or anticonvulsants prescribed for this purpose within 30 days prior to the Screening Visit, or at any time during the screening period
* Any change in the subject's dose or regimen of antispastic agents within the 7 days prior to the Screening Visit, or at any time during the screening period
* Treatment with an investigational drug or approved therapy for investigational use within the 30 days (or 7 half-lives, whichever is longer) prior to the Screening Visit, or at any time during the screening period
* Treatment with 4-AP or 3,4-diaminopyridine (DAP) in any formulation within the 30 days prior to the Screening Visit, or at any time during the screening period
* History of drug or alcohol abuse (as defined by the Investigator) within the 2 years prior to the Screening Visit, or at any time during the screening period
* Female subjects who are currently pregnant or who are considering becoming pregnant while participating in the study. Female subjects of childbearing potential who have a positive pregnancy test at either the Screening Visit or Day 1 may not participate in this study
* Female subjects who are currently breastfeeding
* Inability to comply with study requirements
* Current enrollment in any other drug, biological, device, or clinical study
* Previous participation in this study
* Any other reason, in the opinion of the Investigator, which would disqualify the subject from participation in this study or make the subject unsuitable for enrollment

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in self-assessed walking disability as reported on the Multiple Sclerosis Walking Scale-12 (MSWS-12) | Day 1, up to 24 weeks
Change from baseline in static balance as assessed by Berg Balance Scale (BBS) | Day 1, up to 24 weeks
Change from baseline in dynamic balance as assessed by the Timed Up and Go (TUG) scale) | Day 1, up to 24 weeks
Change from baseline in subjective impression of well-being measured by Multiple Sclerosis Impact Scale-29 (MSIS-29) | Day 1, up to 24 weeks
Change from baseline in subjective impression of well-being measured by Euro Quality of Life-5D (EQ-5D) | Day 1, up to 24 weeks
Participant's global impression of change in walking as reported on the Patient Global Impression of Change Scale (PGIC) | Day 1, up to 24 weeks
Summary of Participants with adverse events (AEs) and serious adverse events (SAEs) | Day 1 Up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (23):
- Belgium (5):
  - Research Site, Ath
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Yvoir
- Canada (5):
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Italy (5):
  - Research Site, Ancona, AN
  - Research Site, Brescia, BS
  - Research Site, Empoli, FI
  - Research Site, Palermo, PA
  - Research Site, Roma, RM
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Sittard-Geleen
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Stockholm
- United Kingdom (4):
  - Research Site, Edgbaston, Birmingham
  - Research Site, Poole, Dorset
  - Research Site, Swansea, Glamorgan
  - Research Site, London

REFERENCES:
- [Background] Hupperts R, Lycke J, Short C, Gasperini C, McNeill M, Medori R, Tofil-Kaluza A, Hovenden M, Mehta LR, Elkins J. Prolonged-release fampridine and walking and balance in MS: randomised controlled MOBILE trial. Mult Scler. 2016 Feb;22(2):212-21. doi: 10.1177/1352458515581436. Epub 2015 Apr 28. PMID 25921050
- See also: EudraCT Tabulated Result — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-000368-90/results